CLINICAL TRIAL: NCT04503785
Title: Esophageal Impedance and Manometry Measurements and Dysphagia Symptom Scoring
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John M. Wo, Director of Motility and Neurogastroenterology Unit, Indiana University
Other Study IDs: 1701721848
Record Dates: First submitted 2018-03-22; First posted 2020-08-07 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia, Esophageal
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dysphagia: Patients with Esophageal dysphagia
  Interventions: Diagnostic Test: Manometry

INTERVENTIONS:
Diagnostic Test: Manometry — Transnasal Esophageal manometry and Endoflip Balloon distensibility
  Other Names: Endoflip

SUMMARY:
Comparison of manometry measurements and EndoFlip Balloon measurements in patients with dysphagia and a known esophageal diagnosis

DETAILED DESCRIPTION:
Gastrointestinal (GI) motility problems are very common in the general population. Dysphagia, difficulty swallowing, is one of the most common issues in gastroenterology. In many patients, esophageal obstruction is not identified despite workup with upper endoscopy or barium swallow x-ray. Patients are often referred to the Motility Laboratory for evaluation of non-obstructive dysphagia. Transnasal esophageal manometry-impedance is a diagnostic test to measure the pressures and coordination of the esophagus during swallowing. The Endolumenal Functional Lumen Imaging Probe (EndoFLIP) is another instrument used to measure the lumen distensibility of the esophagus and pylorus. Both tests are FDA-approved and are currently being used in clinical practice. However, correlation of the results obtained from these tests with clinical syndromes and symptoms is not clearly understood. Furthermore, the relationship between esophageal impedance-manometry and EndoFLIP results has never been defined.

The primary Aim is to develop a registry of patients undergoing esophageal manometry-impedance and Endoflip from the GI Motility Lab at the IU University Hospital

ELIGIBILITY:
Inclusion Criteria:

* All patients who presented to GI Motility Lab at IU University Hospital for esophageal manometry-impedance and/or EndoFLIP

Exclusion Criteria:

* Age <18 yrs old
* Unable to communicate verbally with the staff

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited from patients who were referred by their physicians to the GI Motility Lab at IU University Hospital for esophageal manometry-impedance and/or EndoFLIP
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endoflip parameters for gastroparesis | 5 years
  Compare the distensibility index (mm2/mmHg) of the pylorus at 50 ml distension in patients with postsurgical gastroparesis and compare to patients with idiopathic and diabetic gastroparesis.

SECONDARY OUTCOMES:
Correlation between endoflip parameters and gastric scintigraphy | 5 years
  Correlate distensibility data (cross-sectional area, pressure, distensibility index) with severity of delayed gastric emptying in patients with gastroparesis
Correlation between endoflip parameters and symptom severity | 5 years
  Correlate distensibility data (cross-sectional area, pressure, distensibility index) with severity of gastroparesis symptoms by Patient Assessment GI-Ssymptoms (PAGI-SYM)

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No